CLINICAL TRIAL: NCT05240391
Title: Midodrine Versus Albumin During Large-volume Paracentesis and Its Effect on Paracentesis Induced Circulatory Disturbance in Patients With Acute on Chronic Liver Failure - A Randomized Controlled Trial
Brief Title: Midodrine Versus Albumin for Prevention of Paracentesis Induced Circulatory Disturbance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Dr Mithun Sharma, Director Hepatology and Regenerative Medicine, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AIGHEPAT007
Record Dates: First submitted 2022-01-03; First posted 2022-02-15 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Paracentesis-Induced Circulatory Dysfunction
Keywords: Ascites; Paracentesis-Induced Circulatory Dysfunction; Paracentesis
MeSH Terms: conditions — Ascites | interventions — Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm receiving 20% Human Albumin (Active Comparator): 20% Human albumin given intravenously over 4 hours
  Interventions: Drug: Human Albumin 20%
- Arm receiving Midodrine (Experimental): Tablet Midodrine 2.5 mg - 3 tablets thrice daily orally starting just before paracentesis
  Interventions: Drug: Midodrine Hydrochloride

INTERVENTIONS:
Drug: Midodrine Hydrochloride — Midodrine hydrochloride for PICD prevention
  Arms: Arm receiving Midodrine
Drug: Human Albumin 20% — Human ALbumin 20% for prevention of paracentesis induced circulatory disturbance
  Arms: Arm receiving 20% Human Albumin

SUMMARY:
Paracentesis-induced circulatory disturbance (PICD) is a very common cause of mortality and morbidity in patients undergoing large-volume paracentesis. Albumin is commonly used in decompensated cirrhosis during large-volume paracentesis. However, it may not be cost-effective and has side effects like volume overload and transfusion reactions.

Therefore the investigator proposed to use midodrine which is a drug that increases the mean arterial pressure. The investigators hypothesized that midodrine may be effective in preventing PICD in acute on chronic liver failure patients requiring modest paracentesis. This has already been found to be effective in initial studies in decompensated cirrhosis

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients above 18 years of age who fulfilled Asia Pacific Association of study of liver disease (APASL) criteria for ACLF and required paracentesis for moderate to tense ascites were included in the study.
2. Acute on Chronic Liver Failure (ACLF) was defined as an acute hepatic insult manifesting as jaundice (Serum bilirubin ≥ 5 mg/dL (85 micromole/L) and coagulopathy (INR ≥ 1.5 or prothrombin activity < 40%) complicated within 4 weeks by clinical ascites and/or encephalopathy in a patient with previously diagnosed or undiagnosed chronic liver disease/cirrhosis and is associated with a high 28-day mortality -

Exclusion Criteria:

1. Patients with acute kidney injury defined as serum creatine of > 0.3 mg/dl above the baseline
2. Severe cardiopulmonary disease
3. History of urinary retention
4. Pheochromocytoma
5. Thyrotoxicosis
6. Persistent and excessive supine hypertension define by systolic blood pressure > 150 mm Hg
7. Pregnant patients
8. Unable to give informed consent were excluded from the study -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Prevention of Paracentesis induced circulatory disturbance | Day 6
  Measure the value of plasma renin activity on sixth day after paracentesis

SECONDARY OUTCOMES:
Cost effectiveness of Midodrine versus Albumin | Day 6
  Cost effectiveness of use of Midodrine compared to Albumin
Hepatic Encephalopathy as measured by West-Haven criteria | Day 6
  Hepatic encephalopathy as measured by the West Haven criteria on day 6 in both midodrine and albumin groups
Renal outcome post paracentesis | Day 6
  Serum creatinine, serum sodium and serum potassium values on day 6 after paracentesis

CONTACTS AND LOCATIONS:
Overall Officials: MITHUN SHARMA, MD FACG AGAF, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shrestha DB, Budhathoki P, Sedhai YR, Baniya R, Awal S, Yadav J, Awal L, Davis B, Kashiouris MG, Cable CA. Safety and efficacy of human serum albumin treatment in patients with cirrhotic ascites undergoing paracentesis: A systematic review and meta-analysis. Ann Hepatol. 2021 Dec;26:100547. doi: 10.1016/j.aohep.2021.100547. Epub 2021 Oct 6. PMID 34626828
- [Result] Kulkarni AV, Kumar P, Sharma M, Sowmya TR, Talukdar R, Rao PN, Reddy DN. Pathophysiology and Prevention of Paracentesis-induced Circulatory Dysfunction: A Concise Review. J Clin Transl Hepatol. 2020 Mar 28;8(1):42-48. doi: 10.14218/JCTH.2019.00048. Epub 2020 Mar 26. PMID 32274344
- [Result] Bai M, Han G. Midodrine for paracentesis-induced circulatory dysfunction. J Clin Gastroenterol. 2014 Mar;48(3):300. doi: 10.1097/MCG.0b013e3182a8bfaf. No abstract available. PMID 24100756